CLINICAL TRIAL: NCT00814450
Title: A Prospective, Open-Label, Single-Arm, Single-Center Study Evaluating The Preliminary Safety And Accuracy Of The Actisight™ Needle Guidance System In Patients Undergoing CT-Guided Percutaneous Chest Aspiration And Biopsy
Brief Title: Safety & Accuracy of the ActiSight Needle Guidance System in Percutaneous Chest Aspiration and Biopsy
Acronym: ANGS-PCAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ActiViews Ltd. (Industry)
Responsible Party: Uri Shreter/ Medical Director, Activiews
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ASNG-LFNA-101-IL
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Biopsy
Keywords: Biopsy; Fine needle aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Biopsy needle guidance system (ActiSight™) — The ActiSight system assists in guiding an aspiration or biopsy needle, to a designated point within the body by means of CT visualization.

SUMMARY:
This study is intended to provide clinical data regarding safety and accuracy of the ActiSight™ Needle Guidance System in assisting Chest CT guided biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older at the time of enrollment
* Subjects meeting all medical conditions for percutaneous chest aspiration/biopsy with safe path to lesion between ribs, however, not in the breast area in women or men with gynecomastia
* Single target pulmonary lesion greater than 10 mm in size (diameter) and depth of lesion greater than 40 mm from the skin
* INR <1.3
* Written informed consent to participate in the study
* Ability to comply with the requirements of the study procedures

Exclusion Criteria:

* Fibrous tissue or cyst in access path (not including target lesion)
* Hemophilia, thrombocytopenia, coagulopathy, or other elevated risk for bleeding or abnormal clotting
* Central lesion is located in radius of less than 2 cm from lobar blood vessels and the heart.
* The selected needle path has a safety margin of less than 2 cm from major blood vessels and the heart
* Use of ticlopidine or similar antithrombotic medication
* For subjects taking warfarin or other anticoagulant medication, INR >1.3
* Pulmonary hypertension, heart failure, renal failure, or blood dyscrasia
* Subjects who cannot tolerate mild sedation
* Subjects with FEV1 < 800 mL unless approved by principal investigator following consultation with multidisciplinary team
* Subjects with the following laboratory values, unless approved by hematologist:

  * Platelet count <100,000/mL
  * APTT >39 sec or PT >15 sec
* Pregnancy or lactation
* Patient is unable to comply with requirements of the procedure, i.e. holding breath
* Participation in an investigational trial within 30 days of enrollment
* Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder, or any chronic condition that could, in the opinion of the investigator, of interfering with the conduct of the study.
* Subjects who are uncooperative or cannot follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Frequency of target reached within a radius of 8 mm from the preplanned targeted point as measured on the final CT scan. | Measure evaluated during entire course of study

SECONDARY OUTCOMES:
Number of needle punctures through the skin | Measure evaluated during entire course of study
Number of needle punctures through the pleura | Measure evaluated during entire course of study
Number of CT scans needed | Measure evaluated during entire course of study
Radial distance at target plane at the needle's final position as shown on the ActiSight screen | Measure evaluated during entire course of study
Adverse events following the procedure, including the following:Pneumothorax, Hemoptysis >100 ml, Bleeding, Collapsed lung, Chest drainage, Need for hospitalization | Measure evaluated during entire course of study

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Tiran, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel